CLINICAL TRIAL: NCT07208409
Title: How Small Is Small - Pleurodesis in Small-Bore Chest Tube
Brief Title: Pleurodesis in Small-bore Chest Tube
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW-24-646
Record Dates: First submitted 2025-08-27; First posted 2025-10-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Pleural Effusion, Malignant
Keywords: malignant pleural effusion; pleurodesis; small bore chest tube
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 14 Fr chest tube (Experimental): 14Fr chest tube will be inserted
  Interventions: Device: 14 Fr chest tube
- 12 Fr chest tube (Active Comparator): 12Fr chest tube will be inserted
  Interventions: Device: 12 Fr chest tube
- 8 Fr chest tube (Active Comparator): 8Fr chest tube will be inserted
  Interventions: Device: 8 Fr chest tube

INTERVENTIONS:
Device: 14 Fr chest tube — Chest tube size of 14Fr will be inserted
  Arms: 14 Fr chest tube
Device: 12 Fr chest tube — Chest tube of 12 Fr will be inserted
  Arms: 12 Fr chest tube
Device: 8 Fr chest tube — Chest tube size of 8Fr will be inserted
  Arms: 8 Fr chest tube

SUMMARY:
Malignant pleural effusion (MPE) imposes a high burden on the healthcare system in the Asian Pacific region, as lung and breast cancer are the commonest cancers associated with malignant pleural effusion, as the two commonest cancers in the Asian Pacific region.

While indwelling pleural catheter (IPC), a catheter that is inserted for long-term drainage of pleural fluid, is not commonly used in Asian countries, small-bore chest tubes are increasingly used due to their ease of insertion and causing less pain.

Injecting talc, a chemocal, to promote adhesion of pleura, called talc pleurodesis was an effective method of managing MPE. However, the optimal size of small-bore chest tubes and the feasibility of talc pleurodesis have not been thoroughly investigated.

This randomised controlled trial aims to evaluate the feasibility and success rate of pleurodesis using small-bore chest drains and to examine the outcomes associated with different sizes of these drains, namely 8 Fr, 12 Fr, and 14 Fr, in managing MPE.

The primary outcome is the feasibility of talc pleurodesis with different small-bore chest tubes. Secondary outcomes include the differences in recurrence rates post-pleurodesis between small-bore and ultra-small-bore chest tubes, as well as patient outcomes such as pain scores, SpO2/FiO2 ratios (oxygen saturation/fractional inspired oxygen ratio), and complications.

The sample size will be 60, and the project will be carried out over one year.

The outcome of this study can serve as a reference for managing MPE regarding the feasibility, safety, and efficacy of ultra-small-bore chest tubes worldwide, particularly in the Asia-Pacific region, where IPC is less common.

DETAILED DESCRIPTION:
Chest tubes can be classified as large bore or small-bore base on the size, with commonly ≤14 French (Fr) was defined as small-bore and >14 Fr was defined as large bore. Small-bore chest tubes are increasingly used in malignant pleural effusion (MPE) since it is easier to insert and was reported to have less pain while insertion and in place. However, there is limited evidence and guideline on the use of small-bore chest tube. The size of chest tube for optimal drainage was not mentioned in the British Thoracic Society (BTS) guideline for pleural disease.

Pleurodesis is indicated for MPE or secondary pneumothorax to reduce the recurrent way, and can be performed in surgical or chemical. Different agents are available for chemical pleurodesis, namely talc, minocycline or blood patch. For MPE, talc slurry was shown to be non-inferior than talc poudrage for pleurodesis successful rate, and was shown to be superior than other sclerosant in chemical pleurodesis. For secondary spontaneous pneumothorax, chemical pleurodesis is performed when patient is not a surgical candidate or according to patient's preference. Chemical pleurodesis with talc slurry was shown to have higher efficacy and lower recurrence rate of pneumothorax compared with doxycycline in Asian population.

From the BTS clinical statement on pleural procedures, meta-analyses of studies on different chest tube size for pleurodesis show similar risks of procedure failure with large and small-bore tubes. However, limited evidence was available. The only randomised control trial with adequate sample size found small-bore chest tube was non inferior to large bore chest tube in terms of pleurodesis efficacy. There was a report of use of small-bore chest tube with size 10Fr in MPE, showing response rate of 84.2% post pleurodesis.

The definition of pleurodesis failure in MPE varies. Definition commonly used in previous studies define pleurodesis failure as pleural fluid recurrence in ipsilateral hemithorax requiring further therapeutic pleural intervention, with radiological evidence including chest x-ray (CXR), computed tomography (CT) scan of thorax or transthoracic ultrasound demonstrated same fluid recurrence upon follow up. Partial response was defined as localise effusion that does not progress, cause symptoms or require drainage.

In current practice for chest tube insertion by respiratory team in Queen Mary Hospital, chest tubes with pigtail or seldinger technique are available in size of 8Fr, 12Fr, 14Fr and 18Fr for drainage of pleural effusion or pneumothorax. Pleurodesis, commonly by talc, is performed through chest tubes when clinically indicated.

In this study, we hypothesize that the use of small bore and ultra small bore chest tubes are both effective in managing pleural effusion.

This is a prospective randomised controlled study for patients with MPE who require chest tube insertion. Eligible patients will be randomised into 1:1:1 ratio on 8Fr, 12 Fr or 14 Fr size chest tube. The study will be conducted at Queen Mary Hospital, a tertiary and university-affiliated hospital in Hong Kong.

After study recruitment, chest drain with size according to randomization will be inserted. The baseline characteristics, namely age, sex, underlying malignancy, size of pleural effusion, the patient outcomes including pain score, oxygen saturation, complications including dislodgement, infection, hemothorax, blocked tube and mortality will be analysed between different groups.

For statistical analysis, univariant analysis will be performed first. For categorical factors, including recurrence of pleural effusion or pneumothorax in different groups, Fisher exact test will be performed. Odd ratios will be calculated. Unpaired data on two samples will be performed by Wilcoxon rank sum test. Multivariant logistic regression will then be performed on the effect of different factors on the outcomes. P < 0.05 was taken as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Pleural effusion.
* With clinical indications for pleural drainage and chest drain insertion.
* With anticipated need for pleurodesis e.g. known malignancy, no clinical signs of pleural infection.
* age ≥18 year-old

Exclusion Criteria:

* Pleural effusion not sizable for drainage.
* With clinical suspicion of pleural infection e.g. pleuritic chest pain, fever, ultrasound showed loculated pleural effusion
* Age ≤18 year-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with functional chest tubes after talc pleurodesis in each group | 1 year
  Drainage tube blockage was one of the most common complications for small bore chest tube drainage. While small-bore chest tubes were reported to have similar efficiency for talc pleurodesis, the feasibility of different sizes of small-bore chest tubes i.e. functional chest tubes after talc pleurodesis was not investigated. There is no randomised controlled trial of the feasibility of 8Fr chest tubes compared to other sizes ≤14 Fr. Number of patients with functional chest tube after talc pleurodesis in each group, defined as the chest tube able to drain fluid and air after talc pleurodesis, i.e. not obstructed, is the primary outcome of this study.

CONTACTS AND LOCATIONS:
Overall Officials: King Pui Florence Chan, MD, Principal Investigator — The University of Hong Kong, Queen Mary Hospital
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
According to the current ethics approval protocol, the IPD will be stored anonymously and destroyed 3 years after completion of study.

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Gonnelli F, Hassan W, Bonifazi M, Pinelli V, Bedawi EO, Porcel JM, Rahman NM, Mei F. Malignant pleural effusion: current understanding and therapeutic approach. Respir Res. 2024 Jan 19;25(1):47. doi: 10.1186/s12931-024-02684-7. PMID 38243259
- [Result] Kreisman H, Wolkove N, Finkelstein HS, Cohen C, Margolese R, Frank H. Breast cancer and thoracic metastases: review of 119 patients. Thorax. 1983 Mar;38(3):175-9. doi: 10.1136/thx.38.3.175. PMID 6857580
- [Result] Weichselbaum R, Marck A, Hellman S. Pathogenesis of pleural effusion in carcinoma of the breast. Int J Radiat Oncol Biol Phys. 1977 Sep-Oct;2(9-10):963-5. doi: 10.1016/0360-3016(77)90195-x. No abstract available. PMID 591413